CLINICAL TRIAL: NCT06086535
Title: Intercostal Nerve Cryoanalgesia vs BRILMA Block for Minithoracotomy on Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)324/2022
Record Dates: First submitted 2023-02-18; First posted 2023-10-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Post Operative Pain
Keywords: intercostal nerve cryoanalgesia; BRILMA block; minithoracotomy; cardiac surgery; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BRILMA block: Patients receiving BRILMA blockade. BRILMA blockade will be performed at the end of surgery at the level of the 3rd, 4th and 5th intercostal spaces of the right hemithorax.
  Interventions: Procedure: Intercostal nerve cryoanalgesia vs BRILMA blockade
- Intercostal nerve cryoanalgesia: Patients receiving intercostal nerve cryoanalgesia. The cryoanalgesia technique will be performed by the surgeon before the closure of the minithoracotomy, at the level of the 3rd, 4th and 5th intercostal spaces on the right hemithorax.
  Interventions: Procedure: Intercostal nerve cryoanalgesia vs BRILMA blockade

INTERVENTIONS:
Procedure: Intercostal nerve cryoanalgesia vs BRILMA blockade — For BRILMA block, 0.4 ml/kg of 0.3% ropivacaine will be injected and a catheter will be placed on the 4th intercostal space after surgery. For intercostal nerve cryoanalgesia an external cryogenizer system will be used during surgery

SUMMARY:
Patients undergoing cardiac surgery by minithoracomy present severe acute postoperative pain. Cryoanalgesia of the intercostal nerves and BRILMA block can provide a solution for this postoperative pain. The main aim of this study is to compare the postoperative analgesia provided by BRILMA block and intercostal nerve cryoanalgesia in patients undergoing cardiac surgery by minitoractomia.

DETAILED DESCRIPTION:
Patients undegoing cardiac surgery by minithoracotomy present severe acute postoperative pain. Cryoanalgesia of the intercostal nerves and BRILMA block are performed as techniques of postoperative analgesia of the chest wall, and can provide a solution for this postoperative pain. Both nerve block techniques could have similar effects on postoperative pain control during the first postoperative hours. However, cryoanalgesia of the intercostal nerves may provide a longer duration than that provided by BRILMA block.

Outcomes:

* Compare the postoperative analgesia provided by BRILMA block and intercostal nerve cryoanalgesia in patients undergoing cardiac surgery by minithoracotomy.
* Determine the percentage of patients with neuropathic pain at hospital discharge and 30 days after surgery.

Methods:

Prospective observational study using two analgesic techniques (BRILMA block vs intercostal nerve cryoanalgesia).

Inclusion criteria: patients > 18 years of age, underwent cardiac surgery by minithoracotomy Exclusion criteria: patients <18 years old, patients undergoing cardiac surgery by sternotomy, habitual consumption of analgesics, neurological diseases with deterioration of the level of consciousness and patients with previous neuropathic pain.

Technic: For BRILMA block, 0.4 ml/kg of 0.3% ropivacaine will be injected between the medial aspect of the serratus anterior muscle and the external intercostal muscle (thoraco-dentate space) covering 3 intercostal spaces (3rd, 4th and 5th). A catheter will be placed in the 4th intercostal space that will provide analgesia for the first three postoperative days. The cryoanalgesia technique will be performed by the surgeon before the closure of the minithoracotomy, on the right hemithorax. An external cryogenic system AtriCure CE0123 will be used for use with cryoICE AtriCure 10 cm Cryoablation Probe, CE2797. The cryoprobe will be applied on the lower costal ridge at the level of the 3rd, 4th and 5th intercostal spaces.

Postoperative pain (location and intensity) will be evaluated using a Simple Verbal Scale from 0 (no pain) to 10 (maximum imaginable pain). The need for rescue analgesia will be collected during hospital stay. At 24, 48 and 72 h after surgery and at hospital discharge, the maximum score of pain experienced by the patient (at rest and deep inspiration) will be collected. At hospital discharge, an investigator will evaluate the occurrence of neuropathic pain using the DN-4 scale (Douleur Neuropatique in 4 questions). In addition, the patient will complete these four questions 30 days after surgery and the results will be known by the responsible researcher

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age, underwent cardiac surgery by minithoracotomy
* Cardiac surgery
* Minithoracotomy

Exclusion Criteria:

* <18 years old
* Patients undergoing cardiac surgery by sternotomy
* Patients with regular consumption of analgesics,
* Patients with neurological diseases with altered level of consciousness
* Patients with previous neuropathic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery by minithoracotomy
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | From day of surgery until 30 days after surgery
  Compare the postoperative analgesia provided by BRILMA block and intercostal nerve cryoanalgesia in patients undergoing cardiac surgery by minitoractomia:
  Compare postoperative analgesia provided by BRILMA block and intercostal nerve cryoanalgesia in patients undergoing minithoractomy cardiac surgery:
  1. Determine the location of postoperative pain: in the surgical incision, shoulder, back
  2. Determine the intensity of postoperative pain. Evaluation using simple verbal scale (SVS) of pain: 0 (no pain), 10 (maximum pain) after orotracheal extubation, 24 and 48 hours after surgery and at hospital discharge

SECONDARY OUTCOMES:
Neuropathic pain | 30 days after surgery
  Determine the percentage of patients with neuropathic pain at hospital discharge and 30 days after surgery using the DN-4 scale developed by Bouhassira et al. in 2005

CONTACTS AND LOCATIONS:
Locations (1):
- Susana González Suárez, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khanbhai M, Yap KH, Mohamed S, Dunning J. Is cryoanalgesia effective for post-thoracotomy pain? Interact Cardiovasc Thorac Surg. 2014 Feb;18(2):202-9. doi: 10.1093/icvts/ivt468. Epub 2013 Nov 11. PMID 24218494
- [Result] Saravanan R, Venkatraman R, Karthika U. Comparison of Ultrasound-Guided Modified BRILMA Block with Subcostal Transversus Abdominis Plane Block for Postoperative Analgesia in Laparoscopic Cholecystectomy - A Randomized Controlled Trial. Local Reg Anesth. 2021 Jul 2;14:109-116. doi: 10.2147/LRA.S316320. eCollection 2021. PMID 34239324